CLINICAL TRIAL: NCT01419795
Title: A Phase II Study Investigating Treatment of Post-Allogeneic Transplant Progression or Relapse of CLL/SLL/PLL or NHL With Lenalidomide Alone or With Rituximab
Brief Title: Lenalidomide With or Without Rituximab in Treating Patients With Progressive or Relapsed Chronic Lymphocytic Leukemia, Small Lymphocytic Lymphoma, Prolymphocytic Leukemia, or Non-Hodgkin Lymphoma Previously Treated With Donor Stem Cell Transplant
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohamed Sorror, Principal Investigator, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2467.00; NCI-2011-01703 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA015704 (NIH)
Record Dates: First submitted 2011-08-15; First posted 2011-08-18 (Estimated); Results first posted 2017-03-21 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncutaneous Extranodal Lymphoma; Peripheral T-cell Lymphoma; Prolymphocytic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; T-cell Large Granular Lymphocyte Leukemia; Testicular Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Leukemia, Prolymphocytic; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Leukemia, Large Granular Lymphocytic; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (lenalidomide, rituximab) (Experimental): Patients who have relapsed/progressed within 180 days post-transplant (Cohort 1), beyond day 180 post-transplant (Cohort 2), or within 6 months but were not started within 3 months of relapse, receive lenalidomide PO QD on days 1-28 (patients with CLL/SLL/PLL) or days 1-21 (patients with NHL). Patients in Cohorts 1 and 2 also receive rituximab IV on days 1, 8, 15, and 22 of course 1 and then every two months for courses 3, 5, 7, 9, and 11.
  Interventions: Drug: lenalidomide; Biological: rituximab; Other: pharmacological study; Other: laboratory biomarker analysis
- Arm II (lenalidomide) (Active Comparator): Patients who have relapsed/progressed at any time point post-transplant and who have contraindications, prior severe hypersensitivity reaction to rituximab infusion, to receive rituximab or have CD20 negative disease (Cohort 3) receive lenalidomide as in Arm I.
  Interventions: Drug: lenalidomide; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
  Arms: Arm I (lenalidomide, rituximab)
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving lenalidomide with or without rituximab works in treating patients with progressive or relapsed chronic lymphocytic leukemia (CLL), small lymphocytic lymphoma (SLL), prolymphocytic leukemia (PLL), or non-Hodgkin lymphoma (NHL). Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving lenalidomide together with or without rituximab may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To improve overall survival in patients with relapse of NHL or CLL/SLL/PLL within 180 days after allogeneic hematopoietic cell transplant (HCT).

SECONDARY OBJECTIVES:

I. Rate of response (complete response [CR], partial response [PR], or stable disease [SD]) and time to progression.

II. Grade III-IV toxicity.

III. Incidences of grades II-IV acute graft-versus-host disease (GVHD) and limited or extensive chronic GVHD.

IV. Compare efficacy and safety between the first, second and third cohorts.

V. Laboratory research studies for efficacy and toxicity: blood samples will be stored at baseline, day 7, and day 28 of cycle 1 and day 28 of cycle 3 to investigate:

1. changes in plasma cytokines and peripheral blood lymphocytes in correlation to treatment with lenalidomide;
2. pharmacokinetics of rituximab;
3. donor and host polymorphisms of the FCgamma RIIIa receptor and their impact on disease response and relapse.

OUTLINE: Patients are assigned to 1 of 2 treatment arms.

ARM I: Patients who have relapsed/progressed within 180 days post-transplant (Cohort 1), beyond day 180 post-transplant (Cohort 2), or within 6 months but were not started within 3 months of relapse, receive lenalidomide orally (PO) once daily (QD) on days 1-28 (patients with CLL/SLL/PLL) or days 1-21 (patients with NHL). Patients in Cohorts 1 and 2 also receive rituximab intravenously (IV) on days 1, 8, 15, and 22 of course 1 and then every two months for courses 3, 5, 7, 9, and 11.

ARM II: Patients who have relapsed/progressed at any time point post-transplant and who have contraindications, prior severe hypersensitivity reaction to rituximab infusion, to receive rituximab or have CD20 negative disease (Cohort 3) receive lenalidomide as in Arm I.

Treatment repeats every 28 days for 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 60 days and then every 3 months for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements
* Patients with CLL/SLL/PLL or NHL and who:

  * Met the criteria of relapse or progression after allogeneic HCT according to the HCT protocol or the attending discretion and who,
  * Not responding to appropriate tapering of immunosuppressive medications
* Absolute neutrophil count (ANC) >= 1500/mm^3 or >= 1000/mm^3 if ANC has persistently < 1500/ mm^3 for more than 2 weeks
* Platelet count (transfusion independent) >= 50,000/mm^3 or >= 20,000/mm^3 if platelet count has persistently < 50,000/mm^3 for more than 2 weeks
* Creatinine clearance >= 30ml/min by Cockcroft-Gault formula
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or =< 3 x ULN if total bilirubin has been persistently > 1.5 x ULN for more than 2 weeks
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine transaminase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 3 x ULN or =< 5 x ULN if AST or ALT have been persistently > 3 x ULN for more than 2 weeks
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide; FCBP must also agree to ongoing pregnancy testing; men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist
* Study participants with risk factors for venous thrombo-embolism (VTE), such as previous VTE, cardiac disease, chronic renal insufficiency, and/or poorly controlled diabetes, should be able to comply with some degree of prophylactic anticoagulation using aspirin 81 or 325 mg daily, coumadin, or low molecular weight heparin

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the patient from signing the informed consent form
* Pregnant or breast feeding females; (lactating females must agree not to breast feed while taking lenalidomide)
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Resistance to prior use of lenalidomide, defined as progression on full dose lenalidomide within the first two cycles of therapy
* Concurrent use of other anti-cancer agents or treatments
* Known seropositive for or active viral infection with human immunodeficiency virus
* Karnofsky performance status < 50%
* Active grades III or IV acute graft-versus-host disease (GVHD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sorror, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Started | 3 | 0
Completed | 3 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide) | Total
Number analyzed (Participants) | 3 | 0 | 3
Age, Continuous [Median (Full Range); unit: years] | 57 [48 to 62] |  | 57 [48 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 0 |  | 0
  Unknown or Not Reported | 3 |  | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 3 |  | 3
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Overall Survival of Patients Receiving Lenalidomide With or Without Rituximab in Comparison to Historical Controls Managed by Single or Multiple Chemotherapeutic Agents or Donor Lymphocyte Infusion (DLI) (Cohort 1)
Description: Estimated using the Kaplan-Meier method in all cohorts.
Time Frame: 12 months
Population: Primary objective could not be completed because there were no patients enrolled in the second experimental arm (lenalidomide). Additionally, having only three patients in one arm does not allow for a meaningful comparison to historic controls.
Measure: Number (95% Confidence Interval); unit: survival probability
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
survival probability | 0.33 [0.067 to 1.00] |

2. Secondary Outcome: Rate of Response (CR, PR, or SD) and Time to Progression
Description: Estimated using the Kaplan-Meier method in all cohorts. Assessed at day 100.
Time Frame: Assessed up to 18 months
Population: No participants enrolled in the second arm.
Measure: Number (95% Confidence Interval); unit: progression free survival probability
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
progression free survival probability | 0.67 [0.30 to 1.00] |

3. Secondary Outcome: Grade III-IV Toxicity in Patients Receiving Lenalidomide With or Without Rituximab
Time Frame: Assessed up to 30 days after completion of study treatment
Population: No participants enrolled in the second arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
Participants | 2 |

4. Secondary Outcome: Incidences of Grades II-IV Acute GVHD and Limited or Extensive Chronic GVHD
Time Frame: Assessed up to 30 days after completion of study treatment
Population: No participants enrolled in the second arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
Participants | 0 |

5. Secondary Outcome: Comparison of Rates of Overall Response and Complete Remission Between the First, Second, and Third Cohorts
Time Frame: Assessed up to 18 months
Population: No participants enrolled in the second arm. Not enough participants in first arm to make meaningful comparisons to historic controls.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
Participants | 0 |

6. Secondary Outcome: Changes in Plasma Cytokines and Peripheral Blood Lymphocytes in Correlation to Treatment With Lenalidomide
Time Frame: From baseline to day 28 of course 3
Population: With only 3 participants enrolled to the first arm, meaningful comparisons could not be made and data for this objective was not collected.
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Comparison of Incidences of Adverse Events Between the First, Second, and Third Cohorts
Time Frame: Assessed up to 30 days after completion of study treatment
Population: as for outcome 5
Measure: Number; unit: Number of adverse events
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 3 | 0
Number of adverse events | 7 |

8. Secondary Outcome: Pharmacokinetics of Rituximab: Evaluation of Serum Concentrations and Correlations to Drug Dose and Clinical Responses
Time Frame: Baseline, day 7 and 28 of course 1, and day 28 of course 3
Population: as for outcome 6
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Donor and Host Polymorphisms of the FCgamma RIIIa Receptor and Their Impact on Disease Response and Relapse
Time Frame: Baseline, day 7 and 28 of course 1, and day 28 of course 3
Population: as for outcome 6
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I (Lenalidomide, Rituximab) | Arm II (Lenalidomide)
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Lenalidomide, Rituximab) (N=3) | Arm II (Lenalidomide) (N=0)
Superior vena cava obstruction (Vascular disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Tumor flare syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Rash >50% BSA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes